CLINICAL TRIAL: NCT03008031
Title: Reduced Contrast Administration in Contrast-enhanced Spectral Mammography (CESM)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 162048
Record Dates: First submitted 2016-12-21; First posted 2017-01-02 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Breast Neoplasm; Contrast-enhanced Spectral Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- arm A (40%) (Experimental): Patients randomized in arm A will receive a second CESM exam with 40% of the initial dose of the contrast agent.
  Interventions: Procedure: CESM with a reduced dose of contrast agent
- arm B (60%) (Experimental): Patients randomized in arm A will receive a second CESM exam with 60% of the initial dose of the contrast agent.
  Interventions: Procedure: CESM with a reduced dose of contrast agent
- arm C (80%) (Experimental): Patients randomized in arm A will receive a second CESM exam with 80% of the initial dose of the contrast agent.
  Interventions: Procedure: CESM with a reduced dose of contrast agent

INTERVENTIONS:
Procedure: CESM with a reduced dose of contrast agent

SUMMARY:
The optimal dose of iodine based contrast agents used in contrast-enhanced spectral mammography (CESM) is unknown. If CESM, performed with lower dose of iodine based contrast agent, visualizes a tumor comparable to CESM with regular dose of contrast agent, patients can receive less contrast agent for CESM in future and thereby risking less side effects of the contrast agent.

In order to study whether CESM remains unchanged at smaller amounts of contrast administration, a second CESM exam will be performed within one week of the first with a an alternative amount of contrast, it being either 80%, 60% or 40% of the original contrast dose. The settings of the CESM unit will remain unchanged.

ELIGIBILITY:
Inclusion Criteria:

* Female patient with histopathologically confirmed invasive breast cancer who recently underwent a clinical CESM exam without complications;
* Treated with primary surgery;
* Willing and able to undergo all study procedures;
* Has personally provided written informed consent.
* Age ≥ 18

Exclusion Criteria:

* Pregnancy
* Allergy for any of the ingredients of (Ultravist) contrast agent
* Being unable to give informed consent in person
* History of coronary arterial disease or unstable angina
* Acute or chronic severe renal insufficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Accuracy of maximum tumor size measurements for breast cancer detected with the clinical CESM exam (reference) compared to the (experimental) CESM exams with varying (lower) dose concentrations. | After completion of final patient inclusion (e.g. 1 year)

SECONDARY OUTCOMES:
Enhancement measurements for breast cancer detected with the clinical CESM exam (reference) compared to the (experimental) CESM exams with varying (lower) dose concentrations. | After completion of final patient inclusion (e.g. 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Marc BI Lobbes, MD, PhD, Principal Investigator — Maastricht University Medical Center; Thiemo JA van Nijnatten, MD, PhD — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands